CLINICAL TRIAL: NCT05627050
Title: Online AR Training Platform for the Elderly and Persons With Chronic Diseases at Home
Brief Title: AR Training Platform at Home
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor and Chairman, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020.538
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Stroke; Chronic Disease
MeSH Terms: conditions — Stroke; Chronic Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AR Training System (Experimental): The subjects follow the daily rehabilitation training program designed by clinical and healthcare team. The system will monitor their movement and provide feedbacks to the users. The clinicians/healthcare workers can provide feedbacks and guidance to correct their movements and postures.
  Interventions: Device: An Online Augmented Reality (AR) Training Platform

INTERVENTIONS:
Device: An Online Augmented Reality (AR) Training Platform — The hardware system is based on camera depth sensor and combined with 3D human tracking technology and intelligent technology, to monitor, correct and record the user's whole body movements in real-time, and the users can follow the training program.

SUMMARY:
Video Communications, like ZOOM, have been widely used in the time of this epidemic. But how about to design an AR / VR communication system with coaching from clinician to facilitate training at home in this time of epidemic. Vulnerable individuals at home can interact with the training platform and his/her clinician can provide online training progamme with guidance.

ELIGIBILITY:
Inclusion Criteria:

1. age >=65 years old or suffering from chronic disease;
2. sufficient cognition to follow simple instructions as well as understand the content and purpose of the study MoCA> 21); and
3. Home setting: TV with HDMI input, internet access, and a distance of 1.5m away from TV.

Exclusion Criteria:

1. Any additional medical or psychological condition that would affect their ability to comply with the study protocol, e.g., a significant orthopaedic or chronic pain condition, major post-stroke depression, epilepsy, artificial cardiac pacemaker / joint;
2. Severe shoulder or arm contracture/pain;
3. Severe knee or hip contracture/pain;
4. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | 6-month after the first training
  Fugl-Meyer Assessment for Upper-Extremity the maximum score is 66, divided into 33 items in the form of a 3-point scale (0-2), 0 is cannot perform and 2 performs fully.
  Fugl-Meyer Assessment for Lower-Extremity consists of 34-level cumulative scoring system to examine lower-limb functions of hemiplegic stroke patients quantitatively through a set of lower-limb movement tasks in reflex, flexor/extensor synergy, volitional movement, coordination and speed (Fugl-Meyer, et al., 1975).

SECONDARY OUTCOMES:
The 12-item Short Form Survey | 6-month after the first training
  It is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality-of-life measure.
Barthel Index | 6-month after the first training
  It assesses functional independence, generally in stroke patients.
Berg Balance Scale | 6-month after the first training
  Berg Balance Scale (BBS), consists of 56-level measures to examine balance ability and to predict falling risk with high reliability (ICC=0.98) (Steffen, Hacker & Mollinger, 2002). Stroke patients were assessed based on their performance on 14 simple mobility tasks, including transfer, standing, and reaching
Modified Ashworth Scale | 6-month after the first training
  Modified Ashworth Scale (MAS), consists of 4-level scale to examine joint spasticity based on muscle tone and resistance detected during passive stretching with good inter-rater reliability (ICC =0.85) (Bohannon & Smith, 1987).
Functional Ambulation Category Test | 6-month after the first training
  Functional Ambulatory Category (FAC) is a reliable measurement of independent walking ability on level-ground walking and stair ambulation, which is a good prediction of independent community walking post-stroke (Mehrholz, et al., 2007). FAC consists of 6-level scale: patients with FAC=4 requires supervision in level ground walking, FAC=5 requires supervision only when walking on non-level surface such as stairs.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Kai-yu Tong, PhD, Principal Investigator — Department of Biomedical Engineering, The Chinese University of Hong Kong
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Hong Kong, Hong Kong